CLINICAL TRIAL: NCT03805984
Title: Study to Evaluate the Safety, Tolerability and Immunogenicity of INO-4500 in Healthy Volunteers
Brief Title: Safety, Tolerability and Immunogenicity of INO-4500 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: LSV-001
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Lassa Fever
Keywords: Healthy volunteer
MeSH Terms: conditions — Lassa Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Sponsor will be blinded up to Week 6; at that time the Sponsor will become group-level unblinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- INO-4500 Group A (Experimental): Participants will receive 1 ID injection of 1 mg/dose INO-4500 followed by EP using the CELLECTRA® 2000 device
  Interventions: Drug: INO-4500; Device: CELLECTRA® 2000
- Placebo Comparator Group A (Placebo Comparator): Participants will receive 1 ID injection of 1 mg/dose placebo followed by EP using the CELLECTRA® 2000 device
  Interventions: Drug: Placebo; Device: CELLECTRA® 2000
- INO-4500 Group B (Experimental): Participants will receive 2 ID injections of 1 mg/dose INO-4500 followed by EP using the CELLECTRA® 2000 device
  Interventions: Drug: INO-4500; Device: CELLECTRA® 2000
- Placebo Comparator Group B (Placebo Comparator): Participants will receive 2 ID injections of 1 mg/dose placebo followed by EP using the CELLECTRA® 2000 device
  Interventions: Drug: Placebo; Device: CELLECTRA® 2000

INTERVENTIONS:
Drug: INO-4500 — INO-4500 will be administered ID on Day 0 and Week 4.
  Arms: INO-4500 Group A; INO-4500 Group B
Drug: Placebo — Placebo will be administered ID on Day 0 and Week 4.
  Other Names: SSC-0001
  Arms: Placebo Comparator Group A; Placebo Comparator Group B
Device: CELLECTRA® 2000 — EP using the CELLECTRA® 2000 device will be administered following ID drug administration.

SUMMARY:
This is a randomized and double-blinded within study group, placebo-controlled trial to evaluate the safety, tolerability and immunological profile of INO-4500 administered by intradermal (ID) injection followed by electroporation using the CELLECTRA® 2000 device in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Judged to be healthy by the Investigator on the basis of medical history, physical examination and vital signs performed at Screening;
* Negative tests for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody and Human Immunodeficiency Virus (HIV) antibody;
* Screening electrocardiogram (ECG) deemed by the Investigator as having no clinically significant findings (e.g. Wolff-Parkinson-White syndrome);
* Use of medically effective contraception with a failure rate of < 1% per year when used consistently and correctly from screening until 6 months following last dose or be post-menopausal or be surgically sterile or have a partner who is sterile.

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant or father children within the projected duration of the trial starting with the screening visit until 1 month following last dose;
* Is currently participating in or has participated in a study with an investigational product within 30 days preceding Day 0;
* Previous receipt of an investigational vaccine product for prevention of Lassa Fever;
* Fewer than two acceptable sites available for ID injection and EP considering the deltoid and anterolateral quadriceps muscles;
* Audiometry testing that demonstrates a hearing level threshold of 30 dB or greater for any frequency tested between 250 Hz - 8000 Hz;
* Recent (within 6 months) or planned travel to Lassa-endemic region;
* Current or anticipated concomitant immunosuppressive therapy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Baseline up to Week 48
Percentage of Participants with Injection Site Reactions | Day 0 up to Week 48
Incidence of adverse events of special interest | Baseline up to Week 48

SECONDARY OUTCOMES:
Change from Baseline in Antigen Specific Binding Antibody titers | Day 0 up to Week 48
Change from Baseline in Lassa virus (LASV) Neutralizing Antibodies | Day 0 up to Week 48
Change from Baseline in Interferon-Gamma Response Magnitude | Day 0 up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Mammen Mammen, MD, FACP, FIDSA, Study Director — Inovio Pharmaceuticals
Locations (1):
- The Center for Pharmaceutical Research, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries and all collected IPD will be stripped of identifiers and may be made available upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Anonymous IPD may be shared following or during the publication of summary data. Archival data may be accessed for up to 10 years following the end of the study.
Access Criteria: Those who request the anonymous IPD must provide a plan of study explaining how the data will be used. Requests may be sent to the Central Contact Person. Requests will be reviewed based on the potential for the planned use of the IPD for advancing scientific knowledge and theory.